CLINICAL TRIAL: NCT04313062
Title: Older People Self-caring Through a Comprehensive Model Based on House Calls and Oriented Towards Falling Prevention (PM ACTIVAS)
Brief Title: Falling Prevention Comprehensive Model for Older People Self-caring
Acronym: PMACTIVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Corporación Municipal de Renca, Chile (Unknown); RH Atlantis Healthtech Solutions SPA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ID19I10349
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Accidental Fall; Accident at Home
Keywords: Aged; Accident Prevention; House Calls; Clinical Trial
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive the PM ACTIVAS' intervention model. This intervention will be done by a member of the technical staff (previously trained) at the patient's home (house call). In the house call, the trainee will perform a multidimensional assessment of the patient's falling risks factor (internal and external), deliver a " Falling Prevention Kit " and lastly establish together (with the patient and their family) a plan to change the hazards in their home. The patients will receive a telephone follow-up by the same technical staff member until the final house call, which will be 12 months after the recruiting. Finally, 12 months after recruitment, they will receive a last house call where the trainee will assess with the patient and the family the plan, ask for the " Falls and Events Calendar " given at recruitment (where the older person and/or their family registered every trip or fall during the 12-month period), and conduct the final survey.
  Interventions: Behavioral: Educational Intervention
- Standard care (No Intervention): The control group will receive the standard care from the community health center. They will not receive a telephone follow-up. They will receive a house call 12 months after recruitment by a trainee, who will conduct the final survey and ask for the " Falls and Events Calendar " given at recruitment (where the older person and/or their family registered every trip or fall during the 12-month period). Lastly, they will receive an abbreviated intervention for falling prevention and be given the " Falling Prevention Kit ".

INTERVENTIONS:
Behavioral: Educational Intervention — An educational intervention based on the PM ACTIVAS' model and a " Falling Prevention Kit ", both in a home visit by the trainees. Also, a telephone follow-up and a last house call 12 months after recruiting to assess the changes implemented by the person and their family, to conduct the final survey and to ask for the " Falls and Events Calendar " .
  Other Names: PM ACTIVAS' intervention model
  Arms: Intervention

SUMMARY:
Falls in elderly people are a public health problem and in Chile there's a deficit regarding prevention strategies focused on high functioning older people who live in the community. The aim of the study is to design, implement and evaluate a comprehensive model based on house calls and oriented towards falling prevention (PM ACTIVAS' model). The researchers will perform a clinical trial in a district of Santiago, Chile to evaluate this model. Our hypothesis are that people who received the educational intervention following the PM ACTIVAS' model will: fall less frequently, improve their management on falls risk factors present at home, and have a higher falls risk perception than the control group. The researchers also expect that it will be possible to establish cut off points in a valid and reliable scale to assess the presence of falls risk factors in elderly people.

DETAILED DESCRIPTION:
The comprehensive model PM ACTIVAS uses the house call to make a multidimensional assessment on the patient's falls risks factors (internal and external) and their falls risk perception in order to come up with a plan (together with the patient and their family, if present) to modify the hazards present at the patient's home. Together with a telephone follow-up to support the patient in their plan, it is expected that the patient would have a higher falls risk perception, lower falls risks present at home in order to prevent falling.

In the clinical trial, the sample will comprise of 220 high-functioning elderly people (from 65 to 80 years old) from the area which will be divided in two groups. The intervention group will receive a house call to perform the educational intervention with the PM ACTIVAS' model, while the control group will receive standard care from their health center. The research team will measure their internal and external falls risk factors and their falls risk perception at the beginning and at the end of the study. They will also receive a "Falling Prevention Kit" and a "Fall and Events Calendar" where they have to write every time they fall or trip and the day when it happened. At the end of the study, both groups will receive a house call to measure again their falls risk factors and perceptions in order to analyze if there has been any difference between groups regarding these factors.

ELIGIBILITY:
Inclusion Criteria:

* Older people who has 43 points or more in the elderly functionality test [Examen de Funcionalidad del Adulto Mayor: EFAM] part A test (a chilean validated test that assesses functionality) at recruitment.

Exclusion Criteria:

* Older people whose address does not belong to the health center's territory.
* Older people who have any visual or hearing impairment that hinders effective communication
* Older people with depression or any mild to severe mood disorder stated in their health physical record booklet or drug registry booklet.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Fall frequency | T2 (1 year, final house call)
  Number of falls registered on the " Falls and Events Calendar " in both the control and the intervention group. This calendar is a typical calendar where the patient and/or family have to write the days that the patient fell or tripped. The calendar was given to the patients at recruitment (T0) and have been taught how to register the falls, trips and related events in both groups. The research team will collect the data on the last house call (T2).
Management of external and internal falls risk factors | T0 (recruitment) and T2 (1 year, final house call)
  The research team will measure this with a previously validated checklist, which consists of 41 questions where the patient has to reply yes or no. The questions are related to internal and external falls risk factors. This survey will be applied at the recruitment (T0) and in the last house call (T2) in both control and intervention groups.
Perception on falls risk factors | T0 (recruitment) and T2 (1 year, final house call)
  The researchers will measure the perception that the patient has on falls risk factors in the home setting with a set of drawings where the patient has to identify what they consider as a falls risk factor. The research team will apply this at the recruitment (T0) and in the last house call (T2) in both control and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Bustamante-Troncoso, MNSc RN, Principal Investigator — Profesor Asociado Escuela de Enfermería Pontificia Universidad Católica de Chile; Francisca Márquez-Doren, PhD MNSc RN, Study Director — Profesor Asociado Escuela de Enfermería Pontificia Universidad Católica de Chile
Locations (1):
- Corporación Municipal de Renca, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Marquez-Doren F, Lucchini-Raies C, Alcayaga C, Bustamante C, Gonzalez-Aguero M. Acceptability and feasibility of a comprehensive fall prevention model for independent older adults: A qualitative evaluation. Int J Nurs Stud Adv. 2024 Jun 22;7:100220. doi: 10.1016/j.ijnsa.2024.100220. eCollection 2024 Dec. PMID 39050690